CLINICAL TRIAL: NCT07102368
Title: Generation of Real-world Evidence of Guselkumab in IBD Evaluating Effectiveness, Early Outcomes and Patient Relevant Aspects
Brief Title: A Study to Generate Real-world Evidence of Guselkumab Effectiveness in Inflammatory Bowel Disease in Germany
Acronym: GORGEOUS
Status: Recruiting | Type: Observational
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Other Study IDs: CNTO1959IBD4002; CNTO1959IBD4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease; Colitis, Ulcerative; Crohn's Disease
Keywords: IBD; Ulcerative Colitis; Crohn's Disease; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Pathologic Processes; Inflammatory Bowel Diseases; Colitis, Ulcerative; Ulcer; Guselkumab; Tremfya; Inflammatory
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Pathologic Processes; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Moderate-to-Severe Ulcerative Colitis (UC) or Crohn's Disease (CD): Participants with confirmed diagnosis of moderate-to-severe UC or CD treated with guselkumab as per standard clinical practice will be enrolled. Only data available from clinical routine will be collected in this study. During the observational period, data will be collected at weeks 0 (baseline), 4, 8, 12, 24, 48, 72, and 96, where available as per clinical routine. The respective collection times relate to the first study dose of guselkumab.

SUMMARY:
The purpose of this study is to characterize participants with Crohn's Disease (CD) and Ulcerative Colitis (UC) treated with Guselkumab in a real-world setting, and to assess the clinical effectiveness (how well the treatment works) in the overall population and in different participant subgroups. Furthermore patient-reported outcomes like fatigue, health-related quality of life (HRQoL), sexuality, work productivity and activity as well as treatment satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be eligible for biologic treatment and initiate guselkumab according to the approved indications as described in the current version of the summary of product characteristics
2. Signed informed consent form is available, allowing data collection and source data verification in accordance with local requirements
3. By judgement of the treating physician, the participant is able and willing to complete the patient-reported outcome(s) (PROs) assessments for the duration of the study

Exclusion Criteria:

1. Has a history of more than 4 lines of advanced inflammatory bowel disease (IBD) therapy
2. Has been previously exposed to interleukin (IL)-23 inhibitors. As an exception, participants with history of ustekinumab exposure may be included
3. Has had a colectomy and/or a pouch
4. Is currently enrolled in an interventional clinical study or another non-interventional study from Janssen or Johnson & Johnson (J&J)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with confirmed diagnosis of moderate-to-severe Crohn's disease (CD) or Ulcerative colitis (UC) disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission for Crohn's Disease (CD) as Measured by Harvey-Bradshaw Index (HBI) | Week 48
  Clinical remission for CD is defined as the HBI score less than or equal to (<=) 4. HBI score is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Clinical Remission for Ulcerative Colitis (UC) as Measured by Partial Mayo Score (PMS) | Week 48
  Clinical remission for UC is defined as the PMS score <=2 and a rectal bleeding subscore of 0. Mayo scoring system is used to assess disease severity and treatment effectiveness.

SECONDARY OUTCOMES:
Time to Guselkumab Discontinuation | Up to Week 96
  Time to guselkumab discontinuation (treatment persistency) will be reported.
Change in Stool Frequency Within the First 4 Weeks of Guselkumab Administration | Up to Week 4
  Change in stool frequency for participants will be asked, that is, how many bowel movements they had in last 24 hours, how many of those were very soft or liquid, or how many has occurred during the night.
Change in Rectal Bleeding Within First 4 Weeks of Guselkumab Administration | Up to Week 4
  Change in rectal bleeding for participants will be asked, that is, how severe were the rectal bleedings in the last 24 hours.
Change in Abdominal Pain Within the First 4 Weeks of Guselkumab Administration | Up to Week 4
  Change in abdominal pain for participants will be asked, that is, how severe was the abdominal pain in the last 24 hours.
Change in Bowel Urgency and Nocturnal Bowel Movement (NBM) Within the First 4 Weeks of Guselkumab Administration | Up to Week 4
  Change in bowel urgency and NBM for participants will be asked, that is, how severe were the bowel urgency and NBM in the last 24 hours.
Percentage of Participants Achieving Clinical Response for CD as Measured by HBI | Up to Week 96
  Clinical response for CD is defined as the HBI Score <=4 or a decrease by greater than or equal to (>=) 3. HBI score is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Clinical Response for UC as Measured by PMS | Up to Week 96
  Clinical response for UC is defined as the PMS <4 or >=30% reduction of baseline PMS. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Clinical Remission for CD as Measured by HBI | Up to Week 96
  Clinical remission for CD is defined as the HBI Score <=4. HBI score is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Clinical Remission for UC as Measured by PMS | Up to Week 96
  Clinical remission for UC is defined as the PMS score <=2 and a rectal bleeding subscore of 0. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Corticosteroid-free Clinical Response for CD as Measured by HBI | Up to Week 96
  Corticosteroid-free clinical response for CD is defined as HBI score <=4 or decrease in HBI score >=3 from baseline and no use of steroids for at least 30 days. HBI score is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Corticosteroid-free Clinical Response for UC as Measured by PMS | Up to Week 96
  Corticosteroid-free clinical response for UC is defined as the PMS Score <=4 or >= 30% reduction of baseline and no use of steroids for at least 30 days. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Corticosteroid-free Clinical Remission for CD as Measured by HBI | Up to Week 96
  Corticosteroid-free clinical remission for CD is defined as no use of steroids for at least 30 days and HBI score <=4. HBI score is used to assess disease severity and treatment effectiveness.
Percentage of Participants Achieving Corticosteroid-free Clinical Remission for UC as Measured by PMS | Up to Week 96
  Corticosteroid-free clinical remission for UC is defined as no use of steroids for at least 30 days and PMS <2 and a rectal bleeding subscore of 0. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Percentage of Participants with C-reactive Protein (CRP) Less Than or Equal to 5 milligram/litre (mg/L) | Up to Week 96
  Percentage of participants with CRP level <=5 mg/L, indicating normalization of systemic inflammation will be reported.
Change in CRP Levels | Up to Week 96
  Change in CRP levels will be reported to assess inflammation status.
Percentage of Participants with Fecal Calprotectin (fCAL) Levels Less Than or Equal to 250 microgram/gram (mcg/g) | Up to Week 96
  Percentage of participants with fCal levels <=250 mcg/g will be reported.
Change in fCAL Levels | Up to Week 96
  Change in fCAL levels indicating progression or improvement in inflammation will be reported.
Change in Hemoglobin Levels | Up to Week 96
  Change in hemoglobin levels to assess anemia, measured in gram per deciliter (g/dL) will be reported.
Change in Transferrin Saturation | Up to Week 96
  Serum iron and total iron binding capacity will be combined to report transferrin saturation in percentage (%).
Change from Baseline in Health-related Quality of Life (HRQoL) as Measured by IBD Symptoms | Baseline up to Week 96
  Health related quality of life changes as measured by IBD symptoms (abdominal pain, bowel urgency, nocturnal bowel movements (NBM), rectal bleeding, stool frequency) will be reported. IBD related symptoms changes will be reported by patient diary.
Change from Baseline in General Quality of Life Measured by Short Health Scale (SHS) Score | Baseline up to Week 96
  Quality of life will be assessed by SHS score. SHS is a health related quality of life questionnaire in which the participants rate the disease impact on 4 important aspects of subjective health (symptoms, function, worry, and general well-being). Responses are scored on 100-millimeter (mm) visual analogue scales and presented as individual scores for each of the four questions. The scores are then added for a total score. Total score ranges from 0 (low disease activity) to 100 (high disease activity).
Change from Baseline in IBD-Specific Quality of Life Measured by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Scale Score | Baseline up to Week 96
  SIBDQ is a 10-item instrument developed to assess the participants perception of their health status specifically related to IBD over the past two weeks. The SIBDQ evaluates the following dimensions: psychological well-being (feelings of emotional health and stability), physical well-being (the impact of disease symptoms on physical health), social function (the influence of the disease on social activities and interactions) and digestive function (the effect of gastrointestinal symptoms on daily life). The total score ranges from 10 (worst health) to 70 (best health).
Change from Baseline in Fatigue Measured by Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) Score | Baseline up to Week 96
  FACIT-F is a 13-item questionnaire that evaluates the impact of fatigue on a participants daily life over the past week. It measures various aspects, including: emotional well-being, physical well-being, functional well-being and social/family well-being. The total FACIT-Fatigue score ranges from 0 to 52, with a higher score indicating less fatigue.
Change from Baseline in Treatment Satisfaction Measured by Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) Scores | Baseline up to Week 96
  TSQM-9 is a 9-item general instrument that measures the major dimensions of satisfaction with a medication. The questionnaire consists of 3 domains: effectiveness, convenience and side effects. The scores of each domain range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Change from Baseline in Work Productivity and Activity Impairment Measured by Work Productivity and Activity Impairment (WPAI) Questionnaire | Baseline up to Week 96
  The WPAI consist of four types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. Outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity that is worse outcomes.
Change from Baseline in Sexuality Measured by Intimacy and Sexuality Questionnaire (ISQ)-IBD | Baseline up to Week 96
  The ISQ-IBD is a 5-item questionnaire designed to assess the impact of chronic IBD on participants sexual well-being. Participants are asked to evaluate their situation over the past seven days, with responses tailored to include individuals who may not currently be sexually active. The questionnaire measures various aspects, including: impact of disease on sexual life, satisfaction with physical affection, fear of sexual activity, perceived fear from partner and satisfaction with sexual activity frequency.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 108
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is an important medical event.
Number of Participants with Special Situations | Up to Week 108
  Special Situations include safety events of interest that require reporting for safety evaluation, but are not limited to: drug exposure during pregnancy; exposure to a product from breastfeeding; overdose of a product; suspected abuse/misuse of a product; inadvertent or accidental exposure; any failure of expected pharmacological action; unexpected therapeutic or clinical benefit from use of a product; medication error; suspected transmission of any infectious agent or Off-label use of a product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (1):
- Praxis Fur Gastroenteroligie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No